CLINICAL TRIAL: NCT02987933
Title: The Use of Resting State, fMRI and DTI in the Identification of Chronic Pain Conditions
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Brain Scan Inc. (Industry)
Collaborators: State University of New York at Buffalo (Other)
Responsible Party: Sponsor
Other Study IDs: BSI001
Record Dates: First submitted 2016-12-07; First posted 2016-12-09 (Estimated); Last update posted 2016-12-09 (Estimated); Status verified 2016-12

CONDITIONS: Chronic Pain
Keywords: Chronic Pain; fMRI; DTI
MeSH Terms: conditions — Chronic Pain

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Chronic Pain: Adults, > 6 months duration, daily pain
- Healthy Normals: Age and gender matched controls

SUMMARY:
Resting state fMRI scans of chronic pain sufferers will be compared to those of healthy normals and may be sufficiently different to allow a high level of classification accuracy of whether subjects have chronic pain. In addition, investigators will utilize DTI and a brief activation state using pain rumination to assess whether investigators can reliably find differences between chronic pain sufferers and healthy normals.

DETAILED DESCRIPTION:
Resting state fMRI scans of chronic pain sufferers may be sufficiently different from scans of normal subjects to allow a high level of classification accuracy of whether subjects have chronic pain. In addition, investigators will utilize DTI and a brief activation state using pain rumination to assess whether investigators can reliably find differences between chronic pain sufferers and healthy normals. The analysis will use pattern recognition methods in a leave N out cross validation design. The success of the classifications will be the mean of all the validation runs.

ELIGIBILITY:
Inclusion Criteria:

Daily Pain lasting for more than 6 months. Ages eligible for study are between 20 and 70 years.

Exclusion Criteria:

Adults unable to consent Children, teenagers Pregnant women Prisoners Subjects who do not know English MRI exclusion criteria

Ages: 20 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Adults with daily chronic pain (> 6 months)
Sampling Method: Non-Probability Sample
Enrollment: 40 (Estimated)
Dates: Start 2016-11; Primary Completion 2017-11 (Estimated); Study Completion 2018-01 (Estimated)

PRIMARY OUTCOMES:
Functional brain connectivity | 6 months
  Assessed by fMRI

CONTACTS AND LOCATIONS:
Overall Officials: David S Wack, Ph.D., Principal Investigator — University at Buffalo: SUNY
Locations (1):
- WNY MRI, Buffalo, New York, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Napadow V, LaCount L, Park K, As-Sanie S, Clauw DJ, Harris RE. Intrinsic brain connectivity in fibromyalgia is associated with chronic pain intensity. Arthritis Rheum. 2010 Aug;62(8):2545-55. doi: 10.1002/art.27497. PMID 20506181
- [Background] Kucyi A, Moayedi M, Weissman-Fogel I, Goldberg MB, Freeman BV, Tenenbaum HC, Davis KD. Enhanced medial prefrontal-default mode network functional connectivity in chronic pain and its association with pain rumination. J Neurosci. 2014 Mar 12;34(11):3969-75. doi: 10.1523/JNEUROSCI.5055-13.2014. PMID 24623774
- [Background] Baliki MN, Geha PY, Apkarian AV, Chialvo DR. Beyond feeling: chronic pain hurts the brain, disrupting the default-mode network dynamics. J Neurosci. 2008 Feb 6;28(6):1398-403. doi: 10.1523/JNEUROSCI.4123-07.2008. PMID 18256259
- [Background] Boeckle M, Schrimpf M, Liegl G, Pieh C. Neural correlates of somatoform disorders from a meta-analytic perspective on neuroimaging studies. Neuroimage Clin. 2016 Apr 10;11:606-613. doi: 10.1016/j.nicl.2016.04.001. eCollection 2016. PMID 27182487
- [Background] Tagliazucchi E, Balenzuela P, Fraiman D, Chialvo DR. Brain resting state is disrupted in chronic back pain patients. Neurosci Lett. 2010 Nov 12;485(1):26-31. doi: 10.1016/j.neulet.2010.08.053. Epub 2010 Aug 26. PMID 20800649